CLINICAL TRIAL: NCT05691114
Title: Precise Transplantation of Human Amniotic Epithelial Stem Cells Into Lateral Ventricle for Parkinson's Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai East Hospital (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Principal Investigator, Jingwen WU, Principal Investigator, Shanghai East Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SA-HAES-102
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- hAESCs treatment (Experimental): hAESCs will be administration through Ommaya reservoir implanted into the lateral ventricle.
  The tolerability, safety, and efficacy will be examined of 4 monthly doses of hAESCs for 3 months followed by 2 doses every 3 months in dose escalation through 3 cohorts.
  * Dose A (5×10^7 cells/dose)
  * Dose B (1.0×10^8 cells/dose)
  * Dose C (1.5×10^8 cells/dose).
  Interventions: Biological: hAESCs

INTERVENTIONS:
Biological: hAESCs — human Amniotic Epithelial Stem Cells

SUMMARY:
This is a single-center, single-arm, dose escalation study, to explore the safety, tolerability and efficacy of human amniotic epithelial stem cells (hAESCs) for idiopathic Parkinson's disease (PD).

DETAILED DESCRIPTION:
hAESCs will be administration through the Ommaya reservoir implanted into the lateral ventricle of subjects with idiopathic PD.

This dose escalation will be followed by an exploratory expansion phase in 3 cohorts.

* Dose A (5×10^7 cells/dose)
* Dose B (1.0×10^8 cells/dose)
* Dose C (1.5×10^8 cells/dose).

ELIGIBILITY:
Inclusion Criteria:

1. 40-70 years old, with more than 5 years of idiopathic PD history
2. UPDRS-III off-time scores ≤49
3. MMSE scores ≥24
4. HAMD-17 scores < 25
5. H-Y on-time scores ≤4
6. reactive to levodopa or dopa agonists
7. PD medication dose is stable for more than 2 months
8. no general anesthesia contraindications, no stereotactic surgery contraindications or other conditions that interfere with clinical evaluation
9. no abnormalities affecting cell transplantation by cranial MRI
10. no participation of other clinical trials 3 months before signing the informed consent

Exclusion Criteria:

1. secondary PD or Parkinson's syndrome
2. subcutaneous apomorphine treatment
3. scoring ≥ 2 on UPDRS-I item 2, or ≥ 2 on UPDRS-II item 13; or ≥ 3 on UPDRS-II item14
4. history of intracranial surgery or device implantation, including deep brain stimulation, within 2 years prior to signing informed consent
5. history of seizures or prophylactic application of antiepileptic drugs
6. other serious central nervous system disorders
7. history of stem cell therapy
8. subject who had undergone a major surgery within 3 months and will undergo a major surgery within the next 6 months prior to signing informed consent
9. autoimmune disease or current use of Immunosuppressants
10. subjects with comorbid cardiac disease, for example, but not limited to, ischemic heart disease, congestive heart failure, significant arrhythmias or cardiac conduction block
11. poorly controlled hypertension, diabetes mellitus, or comorbid endocrine system disorders, pulmonary disorders, gastrointestinal system disorders, serious infections, malignancies, etc.
12. positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies, human immunodeficiency virus (HIV) antibodies, or Treponema pallidum antibody
13. abnormalities in liver or kidney function tests, including alanine aminotransferase (ALT), aspartate aminotransferase (AST) is less than 2.5 times the upper limit of normal, blood urea nitrogen (BUN) or creatinine(Cr) are less than 1.5 times the upper limit of normal, or serum albumin < 30.0 g/L
14. abnormalities in hematologic test: coagulation disorders or ongoing anticoagulation therapy; moderate to severe anemia; platelet count < 80 × 10^9/L
15. inability to undergo MRI and positron emission tomography (PET) examinations
16. subject with severe allergies
17. women of childbearing potential (WOCBP) or subject is a man with a WOCBP partner, who are unwilling to take contraception during the trial
18. pregnant or lactating females
19. other conditions deemed by the investigator to be inappropriate for enrollment.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 12 months
  The occurrence of DLT.
Number of participants with adverse event (AE), serious adverse event(SAE) and adverse events of special interest (AESI) | 12 Months
  According to CTCAE V5.0, AE, SAE and AESI evaluated by laboratory examination, measurement of vital signs, physical examination, and subjects' symptoms to detect new abnormalities and/or deterioration of previous conditions.
  AESI is defined as intracranial infection, hemorrhage, rejection, edema, as well as acute allergic reactions and ectopic mass formation associated with the therapy.

SECONDARY OUTCOMES:
Change from baseline in the UPDRS-III (Unified Parkinson's Rating Scale part III/motor part) scores | 12 months
  UPDRS is used for evaluating the impairment and disability associated with PD. It consists of 4 sections: I Mentation, behavior, and mood; II Activities of daily living (ADLs); III Motor; and IV Complications.The UPDRS score ranges from 0 to 199, with higher score indicating greater disability
Change from baseline in the UPDRS off-time total scores | 12 months
  UPDRS is used for evaluating the impairment and disability associated with PD. It consists of 4 sections: I Mentation, behavior, and mood; II Activities of daily living (ADLs); III Motor; and IV Complications.The UPDRS score ranges from 0 to 199, with higher score indicating greater disability
Change from baseline in the UPDRS on-time total scores | 12 months
  UPDRS is used for evaluating the impairment and disability associated with PD. It consists of 4 sections: I Mentation, behavior, and mood; II Activities of daily living (ADLs); III Motor; and IV Complications.The UPDRS score ranges from 0 to 199, with higher score indicating greater disability
Change from baseline in sum of the UPDRS-II and UPDRS-III scores | 12 months
  UPDRS is used for evaluating the impairment and disability associated with PD. It consists of 4 sections: I Mentation, behavior, and mood; II Activities of daily living (ADLs); III Motor; and IV Complications.The UPDRS score ranges from 0 to 199, with higher score indicating greater disability
Changes from baseline in the Parkinson's Disease Questionnaire (PDQ-39) scores | 12 months
  The PDQ-39 is a self-completed questionnaire assessing how often people with Parkinson's experience difficulties across 8 dimensions of daily living with 39 questions . Questions are answered using a 5-point ordinal scoring system: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, 4 = always. Each scores range from 0 = never have difficulty to 100 = always have difficulty.The higher the score, the lower the quality of life of PD patients.
Changes in the Hamilton Depression-17 (HAMD-17) Scale scores | 12 months
  The HAMD-17 Scale is the most widely used scale in clinical evaluation of depression in PD patients. This project takes 8 points as the critical value of depression, and the total score over 35 points is considered as severe depression, more than 20 points is likely to be diagnosed with depression, less than 8 points is not depressed.
Change from baseline in the Parkinson's Disease Sleep Scale (PDSS) scores | 12 months
  The PDSS is a visual analogue scale addressing 15 commonly reported symptoms associated with sleep disturbance overall quality of night's sleep (item 1), sleep onset and maintenance insomnia (items 2 and 3), nocturnal restlessness (items 4 and 5), nocturnal psychosis (items 6 and 7), nocturia (items 8 and 9), nocturnal motor symptoms (items 10-13), sleep refreshment (item 14) and daytime dozing (item 15). Scores range from 0 (poorly or often) to 10 (very good or never), with a total score of <90 indicating sleep disturbance, with higher scores indicating better sleep quality.
Changes from baseline in the Hoehn and Yahr scale (H-Y) | 12 months
  The Hoehn and Yahr scale is used to provide a general estimate of clinical function of PD patients, combining functional deficits (disability) and objective signs (impairment). The Hoehn and Yahr score ranges from 0 to 5, with higher score indicating higher dysfunction of PD patients.
Changes from baseline in the Mini-Mental State Examination (MMSE) | 12 months
  The total score of tne MMSE ranges from 0 to 30, with a higher score indicating better function for Cognitive assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Jingwen Wu, M.D., Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No